CLINICAL TRIAL: NCT00563225
Title: A Multicenter, Non-Comparative, Open, Phase III Study to Evaluate the Efficacy and Safety of Insulin Glargine on Subjects With Type 2 Diabetes Mellitus
Brief Title: 20 Week Bridging Study in Type II DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_3506
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Diabetes Mellitus Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin Glargine — Insulin glargine at the discretion of the investigator Subcutaneous, once daily injection (at bedtime)
  Other Names: Lantus

SUMMARY:
A multicenter, non-comparative, one arm, open, phase III study to evaluate the efficacy and safety of insulin glargine on subjects with Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus diagnosed at least 3 years ago
* Treated concomitantly with insulin once a day and SU over at least 3 months prior to study entry
* Treated with OHA monotherapy over at least 1 year
* HbA1c greater than or equal to 7.5% and less than or equal to 12.0%, at visit 1 (screening visit)
* BMI < 40 kg/m2
* No history of ketonemia
* Women of childbearing potential using the medically approved contraceptive method
* Ability and willingness to perform blood glucose monitoring using a blood glucose meter as per the requirement of protocol

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-10; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To evaluate safety & efficacy of Insulin glargine ( injection at bedtime, once a day) on the changes of HbA1c.

SECONDARY OUTCOMES:
To evaluate the efficacy of Insulin glargine (injection at bedtime, once a day) on the changes of FPG.

CONTACTS AND LOCATIONS:
Overall Officials: Choe Seong Choon, Study Director — Sanofi